CLINICAL TRIAL: NCT04464044
Title: Clinical Performance of a Daily Disposable Toric Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLA306-C003
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Astigmatism
Keywords: Toric contact lens; Daily disposable; Silicone hydrogel contact lens; Axis orientation; Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DDT2 Toric (Experimental): Verofilcon A toric contact lenses worn in both eyes
  Interventions: Device: verofilcon A toric contact lenses

INTERVENTIONS:
Device: verofilcon A toric contact lenses — Daily disposable toric soft contact lenses
  Other Names: DDT2 Toric

SUMMARY:
The purpose of this study is to obtain on-eye clinical performance data to evaluate the stability of axis orientation of DDT2 toric contact lenses in the intended population.

DETAILED DESCRIPTION:
This is a single-visit, non-dispense study where subjects will be exposed to the test lenses for approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an informed consent form;
* Successful wear of spherical or toric soft contact lenses in both eyes, as specified in the protocol;
* Willing to NOT use rewetting/lubricating drops at any time during the study;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any eye condition that would contraindicate contact lens wear, as determined by the Investigator;
* History of eye surgery within the previous 12 months, as specified in the protocol;
* Current or history of dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Percent of lenses with axis orientation within ±30° from the intended axis, 10 minutes after lens insertion | Day 1, 10 minutes after lens insertion
  Axis orientation (orientation of the scribe mark) will be assessed by slit lamp examination and recorded as deviations from intended axis.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No